## **Informed Consent Form**

Title of Project: A Chatbot Intervention for Reducing HPV Vaccine Hesitancy

NCT #: NCT05959564 November 16, 2022

## **CONSENT TO PARTICIPATE**

| Project Title | HPV Vaccine Messaging Survey |
|---|---|
| Purpose of the Study | This research is being conducted by Xiaoli Nan at the University of Maryland, College Park. We are inviting you to participate in this research project because you 1) are at least 18 years old; 2) self-identify as African American; 3) are a custodial parent or caretaker of at least one child ages under 18. The purpose of this research project is to seek community feedback on creating effective HPV (Human Papillomavirus) vaccination messages. |
| Procedures | The procedures completing an online survey. You will answer questions about your attitudes toward childhood vaccines and view one or more HPV vaccine related messages. After that, you will answer questions related to your attitudes toward HPV vaccination, intentions to vaccinate your children, as well as other message response measures. It takes about 10 minutes to complete the survey. Sample questions include "how likely would you be to get your child vaccinated against HPV?" "what's your overall attitude toward HPV vaccination?" |
| Potential Risks and Discomforts | There are no known risks associated with this research. You have the option of not responding to any questions you do not wish to answer. |
| Potential Benefits | There are no direct benefits to you. However, we hope that, in the future, other people might benefit from this study through health communicators' improved understanding of how health messages are being perceived by the target audience, which, in turn, will lead to better health interventions. |
| Confidentiality | Your responses will be confidential. The questionnaires will not contain any questions that ask for information that could be used to identify you. Only approved researchers will have access to the data collected. Hard copy materials will be stored in a locked office. Data collected will be stored in a password-protected computer located in a room with limited access. All research data collected from this study will be stored for 10 years after the study allow the research team to thoroughly analyze the data for research purposes only. The research data will be removed from computer hard disks afterwards. |
| | If we write a report or article about this research project, your identity will be protected to the maximum extent possible. Your information may be shared with representatives of the University of Maryland, College Park or governmental authorities if you or someone else is in danger or if we are required to do so by law. |

| Compensation | You will receive compensation according to the policy of the online survey platform you are using. You will be responsible for any taxes assessed on the compensation. |
|---|---|
| Right to Withdraw and Questions | Your participation in this research is completely voluntary. You may choose not to take part at all. If you decide to participate in this research, you may stop participating at any time. If you decide not to participate in this study or if you stop participating at any time, you will not be penalized or lose any benefits to which you otherwise qualify. |
| | If you decide to stop taking part in the study, if you have questions, concerns, or complaints, or if you need to report an injury related to the research, please contact the investigator: |
| | Xiaoli Nan, Ph.D. Professor, Department of Communication Director, Center for Health and Risk Communication University of Maryland 2102 Skinner Building, 4300 Chapel Ln. College Park, MD 20742 tel: 301-405-0640 fax: 301-314-9471 |
| Participant Rights | If you have questions about your rights as a research participant or wish to report a research-related injury, please contact: |
| | University of Maryland College Park Institutional Review Board Office 1204 Marie Mount Hall College Park, Maryland, 20742 E-mail: irb@umd.edu Telephone: 301-405-0678 |
| | This research has been reviewed according to the University of Maryland, College Park IRB procedures for research involving human subjects. |
| | For more information regarding participant rights, please visit: <a href="https://research.umd.edu/research-resources/research-compliance/institutional-review-board-irb/research-participants">https://research.umd.edu/research-resources/research-compliance/institutional-review-board-irb/research-participants</a> |
| Statement of Consent | By clicking "I agree," you indicate that you are at least 18 years of age; you have read this consent form or have had it read to you; your questions have been answered to your satisfaction and you voluntarily agree to participate in this research study. |
| | If you agree to participate, please click "I agree." |

Page 2 of 2 IRBNet Package: 1960782-1